CLINICAL TRIAL: NCT02824679
Title: Effect of Intravenous Hyoscine Butylbromide Injection on the Course and Duration of First Stage of Labour in Primigavidae
Brief Title: Effect of Intravenous Hyoscine Butylbromide Injection on First Stage Labour in Primigavidae
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ahmed M Maged, MD (Other)
Responsible Party: Sponsor-Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150
Record Dates: First submitted 2016-07-02; First posted 2016-07-07 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Vaginal Delivery
Keywords: Normal labour; Augmentation of labour; Hyoscine butylbromide
MeSH Terms: interventions — Butylscopolammonium Bromide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20mg hyoscine butylbromide (Active Comparator): They received (20mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously
  Interventions: Drug: hyoscine butylbromide; Drug: saline
- 40 mg hyoscine butylbromide (Active Comparator): They received (40mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously
  Interventions: Drug: hyoscine butylbromide
- Saline (Placebo Comparator): They received two ml of normal saline intravenously as a placebo
  Interventions: Drug: saline

INTERVENTIONS:
Drug: hyoscine butylbromide — 20 - 40 mg of hyoscine butylbromide is given intravenously during the first stage of labor
  Arms: 20mg hyoscine butylbromide; 40 mg hyoscine butylbromide
Drug: saline — 0.9%normal saline
  Arms: 20mg hyoscine butylbromide; Saline

SUMMARY:
A case control study conducted on 120 women coming to Cairo University Maternity Hospital .Patients who meet the inclusion criteria were asked to participate in the study and a verbal consent was obtained from each patient. Patients will be divided into three equal groups (A, B, C). A single dose of the drug (placebo or HBB 20mg or HBB 40 mg) will be injected intravenously slowly to groups A, B, C respectively. Labouring mothers will be monitored in bed. Vaginal examination will be conducted every two hours. The duration of the first stage was calculated from the time of cervical dilatation of three to four centimeters in active labour until a fully dilated cervix will be observed

DETAILED DESCRIPTION:
A case control study conducted on 120 women coming to Cairo University Maternity Hospital .Patients who meet the inclusion criteria were asked to participate in the study and a verbal consent was obtained from each patient. Patients will be divided into three equal groups (A, B, C). A single dose of the drug (placebo or HBB 20mg or HBB 40 mg) will be injected intravenously slowly to groups A, B, C respectively. Labouring mothers will be monitored in bed. Vaginal examination will be conducted every two hours. The duration of the first stage was calculated from the time of cervical dilatation of three to four centimeters in active labour until a fully dilated cervix will be observed

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 35 years old
2. Primigravdae.
3. Gestational age between completed 37- 41 weeks + 6 days.
4. Uncomplicated cephalic singleton pregnancy occipto-anterior position.
5. Established spontaneous active labour (defined as the presence of at least three regular uterine contractions over 10 minutes with cervical dilatation three to four centimeters) with cervical effacement not less than 50%.
6. Intact amniotic membranes.

Exclusion Criteria:

1. Multigravidae.
2. Multiple fetus.
3. Malpresentation.
4. Patients with indications of elective caesarean section.
5. Medical conditions associated with pregnancy e.g. preeclampsia, diabetes mellitus.
6. Contraindications for hyoscine butylbromide which include known allergy to hyoscine or other atropinics (e.g., atropine, scopolamine), myasthenia gravis, megacolon or glaucoma.
7. Patients presented to causality with spontaneous rupture of membranes.
8. Spontaneous rupture of membranes during the active phase of first stage of labour.
9. Oxytocin induction or augmentation.
10. Patients who underwent epidural anesthesia or other types of analgesia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
first stage duration | 12 hours after drug intake
  time till cervix become fully dilated

SECONDARY OUTCOMES:
Mode of delivery | 12 hours after drug intake
  Normal vaginal or cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: Yes